CLINICAL TRIAL: NCT04212845
Title: Erector Spinae Plane Block Versus Transforaminal Epidural Injection in Chronic Discogenic Low Back Pain
Brief Title: Erector Spinae Plane Block vs Transforaminal Epidural Injection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Ahmet Murat Yayik, Assistant Professor, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ESPB vs TF
Record Dates: First submitted 2019-12-25; First posted 2019-12-30 (Actual); Last update posted 2020-01-07 (Actual); Status verified 2020-01

CONDITIONS: Discogenic Low Back Pain
MeSH Terms: interventions — Injections; Fluoroscopy; Ultrasonography

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group ESP (Active Comparator): Ultrasound-Guided erector spinae plane block with 30 ml of 0.25% bupivacaine and 8 mg dexamethasone
  Interventions: Drug: Bupivacaine;Dexamethasone Solution for Injection; Device: Ultrasound
- Group TF (Active Comparator): Fluoroscopy-guided transforaminal injection with 4 ml of 0.25% bupivacaine and 8 mg dexamethasone
  Interventions: Drug: Bupivacaine;Dexamethasone Solution for Injection; Device: Fluoroscopy

INTERVENTIONS:
Drug: Bupivacaine;Dexamethasone Solution for Injection — 8 mg Dexamethasone and %0.25 bupivacaine
Device: Fluoroscopy — Fluoroscopy-guided transforaminal injection
  Arms: Group TF
Device: Ultrasound — Ultrasound-guided erector spinae plane block
  Arms: Group ESP

SUMMARY:
Lumbar disc herniation is the main cause of low back pain and radicular leg pain. Steroids administered to the epidural area reduce the inflammatory response and pain by inhibiting the synthesis of proinflammatory agents. Epidural steroid injections are used in the treatment of lumbosacral radicular pain with various techniques including fluoroscopy-guided transforaminal and interlaminar injection.

Ultrasound-guided erector spina plan block (ESPB) was first described in 2016 and has been used for postoperative analgesia in many surgeries including thoracic and lumbar dermatomes. The distribution of local anesthesia in the ESPB from the paravertebral area to the transforaminal and epidural space has been shown in studies.

The aim of this study was to compare the efficacy of ultrasound-guided ESPB and fluoroscopic guided transforaminal epidural steroid injection in chronic discogenic low back pain.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologist's physiologic state I-III patients
* Patients with unilateral radicular pain and low back pain persisting despite medical treatment.

Exclusion Criteria:

* Spinal cord disease or spinal mechanical instability,
* Previous low back surgery,
* More than two levels of lumbar disc hernia,
* Allergic to local anesthetic drugs to be used,
* Use of oral anticoagulants,
* Uncontrolled diabetes mellitus type I and II

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-01-02 (Actual); Primary Completion 2020-06-01 (Estimated); Study Completion 2020-09-01 (Estimated)

PRIMARY OUTCOMES:
Visual analog pain score | Post injection sixth month
  Pain will be evaluated with a Visual Analogue Scale (VAS) score of 0-10 (0= no pain and 10= worst imaginable pain)

SECONDARY OUTCOMES:
Oswestry Disability Index | Post injection first, third and sixth month
  0% -20%: Minimal disability, 21%-40%: Moderate Disability, 41%-60%: Severe Disability, 61%-80%: Crippling back pain, 81%-100%: These patients are either bed-bound or have an exaggeration of their symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Ataturk University, Erzurum, Turkey (Türkiye)

REFERENCES:
- [Background] Celik M, Tulgar S, Ahiskalioglu A, Alper F. Is high volume lumbar erector spinae plane block an alternative to transforaminal epidural injection? Evaluation with MRI. Reg Anesth Pain Med. 2019 Apr 16:rapm-2019-100514. doi: 10.1136/rapm-2019-100514. Online ahead of print. No abstract available. PMID 30992410
- [Background] Makkar JK, Gourav KKP, Jain K, Singh PM, Dhatt SS, Sachdeva N, Bhadada S. Transforaminal Versus Lateral Parasagittal Versus Midline Interlaminar Lumbar Epidural Steroid Injection for Management of Unilateral Radicular Lumbar Pain: A Randomized Double-Blind Trial. Pain Physician. 2019 Nov;22(6):561-573. PMID 31775403